CLINICAL TRIAL: NCT00121940
Title: Guided Care: Integrating High Tech and High Touch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); National Institute on Aging (NIA) (NIH); The John A. Hartford Foundation (Other); The Jacob and Valeria Langeloth Foundation (Other)
Responsible Party: Principal Investigator, Charles Boult, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HS014580-01A1 (AHRQ); HS014580 (Other: NIA- Administrative Supplement); 5R03HS018256 (AHRQ)
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Disease
Keywords: Chronic Disease; Nurses; Caregivers; Support Groups
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided Care (Experimental)
  Interventions: Behavioral: Guided Care
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Guided Care — Specially trained registered nurse (Guided Care Nurse) based in a primary care practice collaborates with two primary care physicians to provide seven services for 40-60 high-risk patients: comprehensive assessment and care planning; "best practices" for chronic conditions; self-management; healthy lifestyles; coordinating care; educating and supporting unpaid caregivers; and accessing community resources.
  Arms: Guided Care

SUMMARY:
The purpose of the study is to evaluate the effect of a Guided Care nurse on the quality of the health and well-being of the frail elderly. A specially trained registered nurse will work closely with 1-3 primary care physicians to provide the most complex older patients (and their unpaid caregivers) with health care that is comprehensive, coordinated, patient-centered, and proactive. The study will evaluate the effects of Guided Care on:

* older persons' physical and mental health, health services utilization, quality of care, self-efficacy, and satisfaction with care;
* older persons' unpaid caregivers' burden; and
* primary care physicians' satisfaction with their care of chronically ill patients.

DETAILED DESCRIPTION:
Health care for older Americans with chronic conditions is often fragmented and provider-centric. In response, a team of investigators at Johns Hopkins University has translated the scientific principles of seven successful innovations into one patient-centered system of care. Supported by evidence-based guidelines and state-of-the-art information technology, "Guided Care" is undergoing a 12-month pilot test in older primary care patients with complex needs. A specially trained Guided Care nurse (GCN), based in a primary care practice, collaborates with two primary care physicians to provide seven services for 40-60 high-risk patients: comprehensive assessment and care planning; "best practices" for chronic conditions; self-management; healthy lifestyles; coordinating care; educating and supporting unpaid caregivers; and accessing community resources.

The proposed multi-site study will measure the effects of Guided Care on the quality and outcomes of care for high-risk older persons, their unpaid caregivers, and their primary care physicians. The panels of 53 physicians in 7 practices will be screened to identify 1350 high-risk older patients. After about 850 have given informed consent and baseline interviews, clusters of 2-5 physicians at each practice site will be randomized to provide either Guided Care or usual care to their consenting patients. Each physician cluster in the Guided Care group will incorporate a GCN into its practice; the physician clusters in the control group will not.

Interviews and queries of administrative databases will provide evaluative data at baseline and at 12-, 24-, and 32-month follow-up intervals. The primary outcome variables are the participants' physical health and mental health (SF-36 Summary Scales) and health services utilization. Secondary outcome variables include: the quality of care; unpaid caregivers' burden; self-rated health; patient satisfaction; and primary care physicians' satisfaction. Intention-to-treat analyses will have 85% power (range of 70-97%) to detect clinically meaningful differences between the two groups.

The study is designed to facilitate the prompt dissemination of Guided Care, if the results of the trial are favorable. A stakeholders' advisory board, representing consumers, providers, delivery systems, insurers, regulators and policy-makers, will inform the operation and evaluation of the study - and it will facilitate the subsequent dissemination of its tools and technology throughout American health care.

ELIGIBILITY:
Inclusion Criteria:

* Over 65
* Insured by KPMAG, USFHP/TRICARE, or Medicare FFS
* High likelihood of use of services in the coming year based on predictive modeling using current year's health care expenses

Exclusion Criteria:

* Moving out of area
* Currently assigned to case manager/in case management program
* Cognitive impairment and no legal representative

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 904 (Actual)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
SF-36 Physical Health Summary Scale | Baseline, 6, 18, and 32 months
SF-36 Mental Health Summary Scale | Baseline, 6, 18, and 32 months
Health Services Utilization | Baseline, 8, 20, and 32 months
  Multiple utilization measures (e.g. hospital admissions, SNF admissions, primary care visits, specialist visits) based on claims data

SECONDARY OUTCOMES:
Perceived Quality of Care | Baseline, 6, 18, and 32 months
  Using Patient Assessment of Chronic Illness Care (PACIC) and Primary Care Assessment Survey (PCAS)
Patient Satisfaction with Care | Baseline, 6, 18, and 32 months
Physician Satisfaction with Care | Baseline, 12, 24, and 36 months
Caregiver Burden | Baseline, 6, and 18 months
  Using Modified Caregiver Strain Index
Self-rated Health | Baseline, 6, 18, and 32 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Boult, MD, MPH, MBA, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Boult C, Reider L, Leff B, Frick KD, Boyd CM, Wolff JL, Frey K, Karm L, Wegener ST, Mroz T, Scharfstein DO. The effect of guided care teams on the use of health services: results from a cluster-randomized controlled trial. Arch Intern Med. 2011 Mar 14;171(5):460-6. doi: 10.1001/archinternmed.2010.540. PMID 21403043